CLINICAL TRIAL: NCT07257328
Title: Comparison of Injectable Platelet-Rich Fibrin (i-PRF) Application and Routine Surgical Extraction on Socket Healing Using a Split-Mouth Technique.
Brief Title: Effect of Injectable Platelet Rich Fibrin (i-PRF) on Extraction Socket Healing: A Split-Mouth Randomized Study.
Acronym: (i-PRF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22-104
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2023-07

CONDITIONS: Wound Healing; Tooth Extraction Site Healing
Keywords: lower third molars; socket healing; i-PRF

STUDY DESIGN:
Intervention Model Description: To reduce inter-individual variability and minimize bias in estimating the treatment effect, the study was designed as a split-mouth trial, with the two treatments randomly assigned to either the right or left side of the dentition.
Who Masked: Outcomes Assessor
Masking Description: The investigators who performed clinical measurements were not involved in the operation and were blinded as to which treatment group the tooth was assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): In the control group, routine surgical extraction will be performed, and the extraction socket will be irrigated with 0.9% physiological saline.
  Interventions: Procedure: Surgical extraction of lower third molars.
- Test group (Experimental): In the test group, routine surgical extraction will be performed, and the extraction socket will be irrigated with i-PRF.
  Interventions: Procedure: Surgical extraction of lower third molars.

INTERVENTIONS:
Procedure: Surgical extraction of lower third molars. — Surgical extraction of lower third molars: Impacted or difficult-to-remove lower wisdom teeth are removed using surgical techniques, involving an incision in the soft tissue and removal of bone.

SUMMARY:
The aim of this study is to compare extraction socket healing (SH) following surgical extraction of lower third molars (LTMs) with and without the application of injectable platelet rich fibrine (i-PRF). A minimum of 32 participants will be included. One mandibular third molar per participant will be randomly assigned to the control group and the contralateral tooth to the test group. SH, gingival recession, and distal periodontal pocket depth of the adjacent second molar will be assessed, and outcomes compared between sides.

DETAILED DESCRIPTION:
Surgical extraction of lower third molars (LTMs) is the most commonly performed procedure in oral and maxillofacial surgery (OMFS). Healing of the extraction socket is a key outcome in oral surgery, as complications in healing may lead to delayed recovery, persistent pain, infection, and adverse events such as dry socket. The aim of this study is to compare extraction socket healing (SH) following surgical extraction of LTMs with and without the application of injectable platelet rich fibrine (i-PRF). For this purpose minimum 32 participants from both sexes will be included to the study. For each participant, one LTM (right or left) will be randomly assigned to the control group and the contralateral tooth to the test group. In the control group, the extraction socket will be irrigated with 0.9% physiological saline solution following standard extraction, whereas in the test group, the socket will be irrigated with i-PRF. SH will be assessed on postoperative days 3 and 14, and at 6 weeks, using the Inflammatory Proliferative Remodeling (IPR) scale and the hydrogen peroxide (H₂O₂) test. Gingival recession and the depth of the periodontal pocket at the distal aspect of the adjacent second molar will be recorded on postoperative days 7 and 14. The outcomes will be compared between the two sides with respect to wound healing.

ELIGIBILITY:
Inclusion Criteria:

Individuals of both sexes Age over 18 years Non-smokers Systemically healthy (ASA I) Requiring surgical extraction of bilateral mandibular third molars

Exclusion Criteria:

Lack of consent to participate Pregnancy Smokers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of socket healing | 6 weeks
  Socket healing of the extracted tooth will be evaluated by using IPR scale which allows to evaluate the healing process according to its biological phases.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)